CLINICAL TRIAL: NCT04000919
Title: The Effects of 5-hydroxytryptophan (5-HTP) and L-3,4-dihydroxyphenylalanine (L-DOPA) Supplementation on Central Nervous System Excitability and Motor Function in Individuals With Spinal Cord Injury
Brief Title: Effects of 5HTP and LDOPA on CNS Excitability After SCI
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI left UofL and intends to reopen study at University of Alberta
Sponsor: Jessica M D'Amico (Other)
Responsible Party: Sponsor-Investigator, Jessica M D'Amico, Assistant Professor, University of Louisville
Organization: University of Louisville (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 18.1268
Record Dates: First submitted 2019-06-19; First posted 2019-06-27 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Carbidopa; Levodopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Both the participant and assessors are blinded to which drug/placebo the participant reviews because all drugs are housed in similar capsules. Only the PI and caregiver will be aware of which drug will be administered for safety purposes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Effects of single-dose of carbidopa (50mg) on CNS excitability (Sham Comparator): Participants will visit the lab and on one of four different occasions they will receive carbidopa only (50 mg). Neurophysiology outcome measures will be obtained at 30, 60, 90, 120 and 150 min post drug-intake.
  Interventions: Drug: Carbidopa
- Effects of single-dose placebo on CNS Excitability (Placebo Comparator): Participants will visit the lab and on one of four different occasions and will receive a placebo. Neurophysiology outcome measures will be obtained at 30, 60, 90, 120 and 150 min post drug-intake.
  Interventions: Drug: Placebo oral tablet
- Effects of single-dose 5HTP/carbidopa on CNS Excitability (Active Comparator): During one of the four occasions participants visit the lab they will receive 5HTP combined with carbidopa (50-200mg HTP/50mg carbidopa). Neurophysiology outcome measures will be obtained at 30, 60, 90, 120 and 150 min post drug-intake.
  Interventions: Drug: 5HTP
- Effects of single-dose L-DOPA/carbidopa on CNS Excitability (Active Comparator): During one of the four occasions participants visit the lab they will receive L-DOPA combined with carbidopa (50-200mg L-DOPA/50mg carbidopa). Neurophysiology outcome measures will be obtained at 30, 60, 90, 120 and 150 min post drug-intake.
  Interventions: Drug: L-DOPA

INTERVENTIONS:
Drug: 5HTP — 5HTP/carbidopa (50-200 mg 5-HTP/50 mg carbidopa)
  Other Names: carbidopa
  Arms: Effects of single-dose 5HTP/carbidopa on CNS Excitability
Drug: L-DOPA — L-DOPA/carbidopa (50-200 mg L-DOPA/50 mg carbidopa)
  Other Names: Sinemet; Carbidopa
  Arms: Effects of single-dose L-DOPA/carbidopa on CNS Excitability
Drug: Placebo oral tablet — Placebo
  Arms: Effects of single-dose placebo on CNS Excitability
Drug: Carbidopa — Carbidopa (50mg)
  Arms: Effects of single-dose of carbidopa (50mg) on CNS excitability

SUMMARY:
This study will examine whether supplementation with the serotonin and dopamine precursors, 5HTP and L-DOPA can alter central nervous system excitability and improve motor function after incomplete and complete spinal cord injuries.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-65 years of age.
* Patients must have suffered a trauma to the spinal cord at least 1 year ago or longer.
* Patients must exhibit some degree of spasticity which can be self-reported (Penn spasm frequency) or if assessed by a physiotherapist, a modified Ashworth spasticity score greater than 1

Exclusion Criteria:

* Individuals with damage to the nervous system other than to the spinal cord
* Pregnant or breastfeeding women
* Alcoholic patients
* Patients with a history of seizures or epilepsy
* Patients with a history of suicidal thoughts or behaviors
* Patients with active or inactive implants including cardiac pacemakers, implantable defibrillators, ocular implants, deep brain stimulators, vagus nerve stimulator, and implanted medication pumps
* Patients with conductive, ferromagnetic or other magnetic-sensitive metals implanted in their head
* Patients with:
* Known or suspected allergy to the medication or the ingredients
* Cardiovascular disease including history of heart attack or heart rhythm irregularities
* Coronary artery disease
* Comatose or depressed states due to CNS depressants
* Endocrine dysfunction
* Blood dyscrasias
* Bone marrow depression
* History of seizures
* Hypocalcemia
* History of stomach ulcers
* Wide-angle glaucoma
* Phenylketonuria

Patients taking:

* Monoamine oxidase inhibitor therapy
* Serotonergic antidepressants: selective serotonin and norepinephrine reuptake inhibitors
* Tricyclic antidepressants
* Any type of serotonergic agonist
* Dopamine D2 receptor antagonists
* Amphetamine
* CNS depressants
* Levodopa
* Lithium
* Anti-hypertensive drugs (Carbidopa and L-DOPA)
* Iron salts
* Metoclopramide
* Phenothiazine medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in corticospinal excitability | Pre drug-intake, 30minutes, 60minutes, 90minutes, 120minutes post drug-intake
  Transcranial magnetic stimulation motor-evoked potentials
Change in motoneuron excitability | Pre drug-intake, 30minutes, 60minutes, 90minutes, 120minutes post drug-intake
  F waves
Change in spinal excitability | Pre drug-intake, 30minutes, 60minutes, 90minutes, 120minutes post drug-intake
  H reflex
Change in spasticity | Pre drug-intake, 30minutes, 60minutes, 90minutes, 120minutes post drug-intake
  Cutaneomuscular reflex
Change in movement performance | Pre drug-intake, 120-150minutes post drug-intake
  Leg cycling

SECONDARY OUTCOMES:
Serum Analysis 5-HIAA | 90-120minutes post drug-intake
  5-HIAA (serum)
Serum Analysis 5-HT | 90-120minutes post drug-intake
  5-HT (serum)
Whole blood analysis 5-HT | 90-120minutes post drug-intake
  5-HT (whole blood)
Serum analysis Cortisol | 90-120minutes post drug-intake
  Cortisol level
Serum and Urine Analysis of dopamine | 90-120min post drug-intake
  catecholamines and homovanillic acid (urine)
Serum Catechloamines | 90-120minutes post drug-intake
  catecholamines and homovanillic acid (urine)
Urine Homovanillic acid | 90-120minutes post drug-intake
  homovanillic acid (urine)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica D'Amico, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Kentucky Spinal Cord Injury Research Centre, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided